CLINICAL TRIAL: NCT01098565
Title: Deep Brain Stimulation Effects: Human Proof-of-Concept Study
Brief Title: Deep Brain Stimulation Effects Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The goal of collecting proof-of-concept information was met through additional modeling studies, new published evidence and information collected from the study
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 1654
Record Dates: First submitted 2010-03-25; First posted 2010-04-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study device arm (Experimental)
  Interventions: Device: Study device HFR0001

INTERVENTIONS:
Device: Study device HFR0001 — Study device will be tested for up to 2 hours prior to chronic device implant.

SUMMARY:
The purpose of this study is to provide proof-of-concept that the test product can perform as intended in an intra-operative setting and the responses to the test product are perceivable in a person. The study will also compare results of the test product to the commercially-available product.

Hypothesis: the test product will elicit successful test results in over 90% of test product.

ELIGIBILITY:
Inclusion Criteria:

* Subject is indicated for Activa® DBS implant for the treatment of Parkinson's disease and scheduled for surgery at the study site.
* Subject is willing to sign the informed consent to participate in the study.
* Subject is 18 years of age or older.
* Subject is a male or non-pregnant female.
* Subject has no factors that would put the subject at an additional risk for intra-operative or postoperative bleeding. This includes underlying disorders of the coagulation cascade (eg, hemophilia), disorders that affect platelet count or function (eg, Von Willebrand's disease), as well as administration of any anti-platelet or anti-coagulant medication in the 7 days prior to surgery, or any history of anticoagulant or aspirin use, that in the view of the neurosurgeon or neurologist would place the subject at an increased risk for intra-operative or postoperative bleeding.

Exclusion Criteria:

* Subject is indicated for DBS for treating a disorder other than Parkinson's disease.
* Subject has any medical contraindications to undergoing DBS surgery, (eg, infection, coagulopathy, or significant cardiac or other medical risk factors for surgery).
* Subject has a history of hemorrhagic stroke.
* Subject has a history of a neurosurgical ablation procedure.
* Subject is currently enrolled in or plans to enroll in any concurrent study that may confound the results of this study, as determined by the investigator or Medtronic.
* Subject has a diagnosis of acute myocardial infarction or cardiac arrest less than or equal to 6 months prior to the screening testing.
* Subject has a history of a seizure disorder
* Subject requires short surgery time due to general health issues, as determined by the investigator.
* Subject is a woman who is pregnant or planning to become pregnant, or a woman of child-bearing potential, who is not using a medically-acceptable method of birth control. Women of child-bearing potential must undergo a pregnancy test, with a clear negative result, no more than 7 days prior to the investigational procedure visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The HFR0001 device can elicit distinct intra-operative responses in subject symptoms. | 9 months
  Responses include testing parameters and symptom effects

SECONDARY OUTCOMES:
Adverse events that occur with the acute implantation and intra-operative testing of the study device. | 9 months.
  Characterization of all adverse events for all subjects from the beginning of the implant procedure through study discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: H. Maximilian Mehdorn, MD, PhD, Principal Investigator — University Clinics Kiel, Department of Neurosurgery
Locations (1):
- Christian Albrechts University of Kiel, Kiel, Germany